CLINICAL TRIAL: NCT01730872
Title: A Single-Center, Double-Masked, Randomized, Placebo-Controlled Evaluation of Prednisolone Sodium Phosphate Ophthalmic Solution, 1% Compared to Placebo in a Modified Conjunctival Allergen Challenge (CAC) Model
Brief Title: Evaluation of Prednisolone in a Modified Conjunctival Allergen Challenge Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-270-0007
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Chronic Allergic Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone (Experimental): Prednisolone Sodium Phosphate Ophthalmic Solution, 1%
  Interventions: Drug: Prednisolone Sodium Phosphate Ophthalmic Solution 1%
- Placebo (Placebo Comparator): Tears Naturale II Ophthalmic Solution, 1%
  Interventions: Drug: Tears Naturale II Ophthalmic Solution

INTERVENTIONS:
Drug: Prednisolone Sodium Phosphate Ophthalmic Solution 1% — One drop in each eye, four times/day for 4 days.
  Arms: Prednisolone
Drug: Tears Naturale II Ophthalmic Solution — one drop in each eye, four times/ day (QID) for 4 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the modified Conjunctival Allergen Challenge (CAC) and observe how the produced allergic inflammation reacts to treatment with a proven ocular anti-inflammatory medication,

Prednisolone, assessed by the following measures:

Chronic Allergic Inflammation assessed using confocal microscopy Ocular itching Conjunctival redness

DETAILED DESCRIPTION:
Prospective, single center, randomized, double-masked, placebo controlled study. Subjects will be randomized to one of the following treatment arms to dose four times per day (QID) for 4 days between Visits 3 and 4.

Prednisolone phosphate Tears Naturale II Ophthalmic Solution (Placebo)

Duration:

Approximately 2 weeks

Controls:

Artificial Tears (Tears Naturale® II)

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age & either sex, any race
* Willing and able to follow all instructions
* Positive history of ocular allergies
* Reproducible positive ocular allergic reaction induced by conjunctival allergen challenge

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy or lactating
* Use of disallowed medications
* Have ocular infections, or ocular conditions that could affect study parameters
* Have moderate to severe dry eye
* Have used an investigational drug or device within 30 days of start of study
* Female that is currently pregnant, planning a pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Massachusetts Medical Society, Alpha Omega Alpha Honor Society, American Academy of Ophthalmology
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Subjects received CAC using saline instead of allergen
Period: Overall Study
Arm/Group | Prednisolone | Placebo | Control
Started | 8 | 5 | 3
Full Analysis Set | 8 | 4 (1 subject did not complete the last post-CAE measurement on Day 6 and was excluded from the FAS) | 0
Completed | 8 | 5 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Saline: A group of three allergic subjects will be challenged with saline only to evaluate the impact of confocal microscopy on ocular signs and symptoms in the absence of allergic challenge. These five subjects will receive placebo in an open label fashion and will not require randomization.
- Total: Total of all reporting groups
Arm/Group | Prednisolone | Placebo | Saline | Total
Number analyzed (Participants) | 8 | 5 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.75 (1.461897) | 37.2 (1.830301) | 39.33 (0.905539) | 39.88 (0.0707107)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 5 | 3 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 4 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Inflammation Change From Baseline to Day 6
Description: Ocular inflammation was measured by a masked clinician on a 4-point scale 90 minutes after the conjunctival allergen challenge (CAC) . 0 = best (little to no inflammation), 4 = worst (most inflammation).
Time Frame: 90 minutes post CAC
Population: The per-protocol (PP) population will comprise all subjects in the ITT population without protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 8 | 4
score on a scale | -1.2 (0.78) | -0.19 (0.43)

2. Secondary Outcome: Ocular Itching Change From Baseline to Day 6
Description: Ocular itching was measured by subject on a scale of 0 to 4 where 0 = no itching and 4 = worst itching. This measurement was taken 7 minutes post CAC
Time Frame: 7 minutes post-CAC
Population: The per-protocol (PP) population will comprise all subjects in the ITT population without protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 8 | 4
score on a scale | -1.1 (1.30) | -1.0 (1.29)

3. Secondary Outcome: Ocular Redness Change From Baseline to Day 6
Description: Ocular redness was measured by the investigator on a 4-point scale 7 minutes post-CAC. 0 = best (no redness), 4 = worst (most redness).
Time Frame: 7 minutes post-CAC
Population: The per-protocol (PP) population will comprise all subjects in the ITT population without protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 8 | 4
score on a scale | -1.1 (1.38) | 0.31 (1.01)

ADVERSE EVENTS:
Time Frame: AEs were collected from the signing of the informed consent form to the end of the study (approximately 2 weeks).
Groups:
- Saline: A group of five allergic subjects will be challenged with saline only to evaluate the impact of confocal microscopy on ocular signs and symptoms in the absence of allergic challenge. These five subjects will receive placebo in an open label fashion and will not require randomization.
Arm/Group | Prednisolone | Placebo | Saline
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 2/8 | 1/5 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=8) | Placebo (N=5) | Saline (N=3)
peri-ocular lid redness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
lower leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
endothelial pigment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No